CLINICAL TRIAL: NCT06086678
Title: Improvement of Pulmonary Function in Hemiplegic Cerebral Palsied Children by Using Hydrotherapy and Aerobic Exercises
Brief Title: Effect of Hydrotherapy Versus Aerobic Exercise on Pulmonary Function on Hemiplegic Cerebral Palsied Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ragaee Saeed Mahmoud, Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004140
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: To Compare the Effectiveness of Hydrotherapy Versus Aerobic Exercise on Pulmonary Function in Hemiplegic Children With Cerebral Palsy
Keywords: Aerobic exercise; Cerebral palsy; Children; Hemiplegia; Pulmonary function
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia | interventions — Physical Therapy Modalities; Hydrotherapy; Exercise

STUDY DESIGN:
Intervention Model Description: random
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional physical therapy group (Experimental): Strengthening exercises, stretching exercises for the weak and tightened muscles respectively, facilitation of equilibrium and protective reactions and breathing exercises in form of Deep breathing, Diaphragmatic breathing and Pursed lip breathing exercises
  Interventions: Other: Conventional physical therapy
- Hydrotherapy and conventional physical therapy group (Experimental): Strengthening exercises, stretching exercises for the weak and tightened muscles respectively, facilitation of equilibrium and protective reactions and breathing exercises in form of Deep breathing, Diaphragmatic breathing and Pursed lip breathing exercises in addition to hydrotherapy
  Interventions: Other: Conventional physical therapy; Other: Hydrotherapy
- Aerobic exercise and conventional physical therapy group (Experimental): Strengthening exercises, stretching exercises for the weak and tightened muscles respectively, facilitation of equilibrium and protective reactions and breathing exercises in form of Deep breathing, Diaphragmatic breathing and Pursed lip breathing exercises in addition to aerobic exercise
  Interventions: Other: Conventional physical therapy; Other: Aerobic exercise

INTERVENTIONS:
Other: Conventional physical therapy — 1. Deep breathing exercise.
  2. Diaphragmatic breathing exercise.
  3. Pursed lip breathing exercise.
  Other Names: Physical therapy
Other: Hydrotherapy — 1. Water walking exercise.
  2. Forward lunges exercise.
  3. Single leg balance exercise.
  4. Side stepping exercise.
  5. Push ups exercise.
  6. Standing knee lifts exercise.
  Other Names: Physical therapy
  Arms: Hydrotherapy and conventional physical therapy group
Other: Aerobic exercise — Aerobic exercise in form of treadmill training when each child was standing on the treadmill, should be ensure that this standing in an upright position, and according to each child, the therapist corrected the height of the handrails. Ask the child to keep looking forwards along the walking on the treadmill aiming to encourage the setting of walking free. The treadmill training would be completed for each child when the child completes three stages in 1-min training cycles. First stage: the child grasped on to the rails with both hands in first 15 s of every 1-min. Second stage: the child grasped on to the railings with one hand in the second 15 s. And final stage: the child didn't grasp on to the railings in last 30 s. Every child performed this procedure twenty times
  Other Names: Physical therapy
  Arms: Aerobic exercise and conventional physical therapy group

SUMMARY:
Cerebral palsy (CP) is the most common motor disability in childhood. Respiratory muscle weakness and a low upper to lower chest diameter ratio are common respiratory dysfunction manifestations in those children which negatively affect their quality of life..

DETAILED DESCRIPTION:
Objective: To compare the effectiveness of hydrotherapy versus aerobic exercise on pulmonary function in hemiplegic children with cerebral palsy. Methods: Sixty hemiplegic children (both genders) took part in this research, they were between the ages of 8 to 16, moreover, they were split equally between three groups (A, B and C). The three groups participated in the same conventional physical therapy, group (A) received conventional physical therapy only, group (B) received hydrotherapy, while group (C) received aerobic exercise. Pulmonary function tests are measured by Six-minute walk test (6-MWT) and Spirometer to measure Forced vital capacity (FVC), Forced expiratory volume in the first second (FEV1) as well as FEV1/FVC ratio for all children before the beginning and after the end of this study, the treatment program was applied three sessions per week for 12 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ages ranged from 8 to 16 years.
* Belonged to levels I to II of the Gross Motor Function Classification System (GMFCS).
* Spasticity ranged from grade 1 to grade 1+ according to Modified Ashwarth Scale. - Able to walk, no impairment of sensation or other neurological or psychological problems.
* Clinically and medically stable and able to understand and follow the instructions

Exclusion Criteria:

i) Visual and/or auditory defects. ii) Significant shortening and/or deformity of lower extremities. iii) Other neurological problems that affect balance or mentality (e.g. epilepsy) iv) Advanced radiographic alterations comprise (bone destruction, bony ankylosis, knee joint sublaxation as well as epiphysial fracture).

v) Lower extremity skeletal abnormalities (whether congenital or acquired). vi) Cardiopulmonary dysfunction.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | 12 consecutive weeks
  Pulmonary function test
Pulmonary function tests Forced expiratory volume in the first second (FEV1) | 12 consecutive weeks
  Pulmonary function test
FEV1/FVC ratio | 12 consecutive weeks
  Pulmonary function test

SECONDARY OUTCOMES:
Six-minute walk test (6-MWT) | 12 consecutive weeks
  It assesses exercise capacity objectively and determine prognosis in many respiratory (such as COPD, idiopathic pulmonary fibrosis, and pulmonary hypertension) and non-respiratory conditions (such as heart failure)

CONTACTS AND LOCATIONS:
Locations (1):
- Ragaee Saeed Mahmoud, Giza, Faisal, Egypt

IPD SHARING:
Plan to Share IPD: No